CLINICAL TRIAL: NCT04138927
Title: A Phase 3 Open Label Extension Study of Fostamatinib Disodium in the Treatment of Warm Antibody Autoimmune Hemolytic Anemia
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-935788-058
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-07

CONDITIONS: Warm Antibody Autoimmune Hemolytic Anemia
Keywords: wAIHA; Warm Antibody Autoimmune Hemolytic Anemia; Warm Autoimmune Hemolytic Anemia
MeSH Terms: interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fostamatinib (Experimental): Subjects who at any time during the C-935788-057 study achieved a hemoglobin response will continue at their dose and regimen from the Week 22 visit in the C-935788-057 study.
  All other subjects who enter the extension study will initially receive fostamatinib 100 mg PO bid. Starting at Week 4, the initial fostamatinib dose of 100 mg PO bid will be increased to fostamatinib 150 mg PO bid if subjects have adequately tolerated the study drug, based on the Investigator's judgment.
  Interventions: Drug: Fostamatinib disodium

INTERVENTIONS:
Drug: Fostamatinib disodium — Fostamatinib is supplied in two (2) dosage strengths: 100 mg and 150 mg.
  Other Names: R935788; Fostamatinib

SUMMARY:
The primary objective of this study is:

• To evaluate the long-term safety of fostamatinib in subjects with warm antibody autoimmune hemolytic anemia (wAIHA).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be willing and able to give written informed consent by signing an IRB approved Informed Consent Form prior to undergoing any study-specific procedures.
2. Subject must have completed all 24 weeks of participation in the study C-935788-057.

Exclusion Criteria:

1. Any subject who discontinued participation in Study C-935788-057 prior to Week 24.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 104 weeks
  Incidence, frequency, seriousness, and severity of adverse events that occurred during the current study
Blood Pressure | 104 weeks
  Change from baseline in blood pressure over time
Absolute Neutrophil Count (ANC) | 104 weeks
  Change from baseline in absolute neutrophil count (ANC) over time

SECONDARY OUTCOMES:
Achievement of Durable Hemoglobin Response | 24 weeks
Total Duration of Response | During the Intervention period up to 104 weeks
Corticosteroid dose | During the Intervention period up to 104 weeks
  Net cumulative change from Baseline in corticosteroid dose

CONTACTS AND LOCATIONS:
Locations (37):
- United States (8):
  - University of Southern California - Janice and Robert Hall Clinical Trials Biospecimen Laboratory, Los Angeles, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - American Oncology Network Vista Oncology Division, Olympia, Washington
  - University of Washington, Seattle, Washington
- Australia (2):
  - Princess Alexandra Hospital - Cancer Trials Unit, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Hanusch-Krankenhaus, Vienna
  - Universitätsklinik f. Innere Medizin I - Klin. Abt. f. Hämatologie u. Hämostaseologie, Vienna
- Belarus (2):
  - Vitebsk Regional Clinical Hospital, Vitebsk
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- AZ Nikolaas, Sint-Niklaas, Belgium
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv, Clinic of Medical oncology, Pleven
  - University Multiprofile Hospital for Active Treatment Sv. Ivan Rilski EAD, Varna, Clinic of Clinical Haematology, Sofia
  - Specialized Hospital for Active Treatment of Hematological Disease EAD,, Sofia
- Czechia (2):
  - Fakultni nemocnice Brno Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Ostrava Klinika hematoonkologie, Ostrava
- CHU de Bordeaux - GH Sud- Hôpital Haut Lévêque Service Médecine Interne et Maladies Infectieuses, Pessac, France
- Georgia (2):
  - LTD Multiprofile Clinic Consilium Medulla, Tbilisi
  - M. Zodelava Hematology Centre, Tbilisi, Tbilisi
- Universitätsklinikum Essen, Essen, Germany
- Italy (3):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, UO Ematologia, Milan
  - Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico di Milano - UO Ematologia, Milan
  - SCDU Ematologia AOU "Maggiore della Carità", Novara
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Haukeland University Hospital, Bergen, Norway
- Russia (2):
  - National Research Center for Hematology, Moscow
  - State Budgetary Healthcare Institution Oncology Dispensary No. 2 of the Ministry of Health of the Krasnodar Territory, Sochi
- Clinical Centre of Vojvodina, Clinic for Hematology, Novi Sad, Serbia
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
- Ukraine (2):
  - City Clinical Hospital № 4, Hematology Center, Dnipro
  - Kyiv City Clinical Hospital №9, hematology department №1, Kyiv
- Roald Dahl Haemostasis and Thrombosis Centre, Royal Liverpool University Hospital, Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No